CLINICAL TRIAL: NCT01450189
Title: Acute HIV Infection - A Key Link for Transmission Prevention: A Randomized Pilot Study
Brief Title: A Key Link for Transmission Prevention
Acronym: MP3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-0815; CID 1002 (Other: UNC Chapel Hill)
Record Dates: First submitted 2011-09-18; First posted 2011-10-12 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2016-11

CONDITIONS: HIV
Keywords: Acute HIV; Transmission Prevention; Randomized Pilot study
MeSH Terms: interventions — Raltegravir Potassium; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Counseling Arm (Active Comparator): The SC arm consists of a single session of standard HIV prevention messages during HIV post-test counseling. The counseling will be comparable to that given to persons with established HIV infection with supplemental information regarding the acute stage of their infection.
  Interventions: Behavioral: Standard HIV prevention messages
- Behavioral Intervention Arm only (Active Comparator): Behavior- BI: Information-Motivation-Behavioral Skills Model the Information-Motivation-Behavioral Skills (IMB) Model. The 5 sessions are designed to provide participants with the information, motivation, and skills needed to abstain or practice protected sex during the brief acute HIV period, as well as plan for long-term behavioral risk reduction.
  Interventions: Behavioral: Standard HIV prevention messages; Behavioral: BI: Information-Motivation-Behavioral Skills Model
- Behavioral Intervention plus ARV (Active Comparator): The BIA arm consists of the behavioral intervention plus antiretroviral drugs (ARVs) with raltegravir (400 mg twice daily) and fixed dose combination (FDC) emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) (200/300 mg daily) orally for 12 weeks.
  Interventions: Behavioral: Standard HIV prevention messages; Behavioral: BI: Information-Motivation-Behavioral Skills Model; Drug: Raltegravir; Drug: emtricitabine/tenofovir disoproxil fumarate

INTERVENTIONS:
Behavioral: Standard HIV prevention messages — A single session of standard HIV prevention messages during HIV post-test counseling with supplemental information regarding the acute stage of their infection.
Behavioral: BI: Information-Motivation-Behavioral Skills Model — The behavioral intervention consists of five counselor-delivered sessions based on the Information-Motivation-Behavioral Skills (IMB) Model. The sessions are designed to provide participants with the information, motivation, and skills needed to abstain or practice protected sex during the brief acute HIV period, as well as plan for long-term behavioral risk reduction.
  Arms: Behavioral Intervention Arm only; Behavioral Intervention plus ARV
Drug: Raltegravir — raltegravir (400 mg) administered orally twice daily for 12 weeks
  Other Names: Isentress, RAL
  Arms: Behavioral Intervention plus ARV
Drug: emtricitabine/tenofovir disoproxil fumarate — emtricitabine/tenofovir (200/300 mg daily) in a fixed dose combination administered orally for 12 weeks
  Other Names: Truvada, FTC/TDF
  Arms: Behavioral Intervention plus ARV

SUMMARY:
This pilot study will assess the feasibility for the potential public health benefit of behavioral and antiretroviral interventions during acute HIV infection.

Central Hypothesis The investigators hypothesize that delivering behavioral and antiretroviral interventions to acutely infected persons will reduce onward transmission.

DETAILED DESCRIPTION:
The HIV epidemic in sub-Saharan Africa is severe and continues to grow. In urban areas of Malawi, 19% of pregnant women seeking antenatal care and 15.6% of Malawians aged 15-49 years were infected with HIV in 2007. Prevention interventions that prevent onward transmission of HIV are urgently needed.

Persons with acute HIV infection (AHI) may be responsible for a substantial proportion of onward transmission of HIV infection. AHI is characterized by unfettered replication of HIV in a "ramp up viremia". The high concentration of HIV in blood and genital secretions remains elevated for up to 10-12 weeks before it declines to the levels observed in established infection. These high levels of HIV shedding in the genital tract are likely to produce very efficient sexual transmission and the proportion of virions that are infectious may be substantially higher during acute compared to chronic infection. Consequently, the probability of transmission during unprotected intercourse for those with AHI is very high. Identifying persons with AHI and intervening to reduce onward transmission represents a tantalizing, but unproven, opportunity for HIV prevention.

To have maximal impact, a prevention program targeting AHI must identify a substantial number of acutely infected persons and intervene quickly to minimize onward transmission. An effective immediate intervention would require behavioral modification to limit sexual partners and unprotected sex acts, and a biological intervention to reduce infectious viral burden in genital secretions. This is the first study to pilot a combined behavioral and biomedical intervention in individuals with AHI to reduce onward transmission of HIV.

ELIGIBILITY:
Inclusion Criteria:

Primary participants:

* Acute HIV-1 infection
* Men and women age greater than/= 18 years.
* Intention to remain in the Lilongwe area for the duration of the study.
* Ability and willingness of participant to provide informed consent.
* Willingness to provide contact/locator information, be contacted, and asked to return for AHI results.

Partner Participants:

* Referred by a primary participant and present with a referral card.
* Had vaginal or anal sex with a primary participant within 12 weeks prior to that primary participant's enrolling
* Men and women age greater than/=18 years.
* remain in the Lilongwe area for the duration of the study.
* Ability and willingness of participant to provide informed consent.

Exclusion Criteria:

Primary Participants:

* HIV infection based on two positive HIV antibody rapid tests at the time of screening.
* HIV-negative based on one or more antibody rapid test and an HIV RNA PCR test.
* Serious illness, including tuberculosis or opportunistic infection, requiring systemic treatment and/or hospitalization.
* Active drug or alcohol use or dependence.
* Current imprisonment or involuntary incarceration.
* Any other condition that in the opinion of the study investigator would compromise the safety of the study participant or study staff, or would prevent proper conduct of the study.

Partner Participants:

* Active drug or alcohol use or dependence.
* Current imprisonment or involuntary incarceration in a medical facility for psychiatric or physical illness.

Exclusion for Receipt of Antiretroviral Drugs in the BIA Arm

Note:A key component of this pilot study is to estimate the potential effect of ARVs during acute infection when applied on a large population scale.In effect, this pilot study should be viewed as a pilot for an effectiveness trial. Consequently, we will randomize all eligible participants to one of the three arms. If, however, persons should not receive ARVs for a variety of medically-related reasons, these persons will remain in the BIA arm, but will not receive ARVs. Women who are of reproductive potential but who refuse to use at least one form of contraception (see below), will remain in the BIA arm but will not receive ARVs. Similarly, persons randomized to the BI arm who do not attend all sessions will remain in the BI arm.

Persons randomized to BIA with any of the following conditions will be excluded from receiving ARVs, but will remain in the BIA group for purposes of analysis.

* Laboratory values obtained at Day 0 prior to initiating ARVs at a subsequent visit
* Absolute neutrophil count <300/mm3
* Hemoglobin <8.0 g/dL
* Platelet count <40,000/mm3
* Aspartate aminotransferase, alanine aminotransferase, and alkaline phosphatase > 5 x upper limit of normal (ULN)
* Total bilirubin >2.5 x ULN
* Creatinine Clearance (CrCl) <60 mL/min
* Hepatitis B surface antigen positivity
* Positive serum or urine pregnancy test at Day 0.
* Breastfeeding
* Refusal to use at least one method of contraception, if a woman is of reproductive potential.

Acceptable forms of contraception include: condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, intrauterine device (IUD), or a hormonal-based contraceptive.

Women not meeting the reproductive potential criteria above may receive the study drugs without using contraception.

* Known allergy/sensitivity or any hypersensitivity to components of study drug(s) or their formulation.
* Requirement for any current medications that are prohibited with any study drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C Miller, MD, PhD, MPH, Study Chair — University of North Carolina, Chapel Hill; Audrey Pettifor, PhD, MPH, Study Chair — University of North Carolina, Chapel Hill; Sam Phiri, PhD, MSc, Principal Investigator — Kamuzu Central Hospital
Locations (2):
- Malawi (2):
  - Lighthouse Trust, Kamuzu Central Hospital, Lilongwe
  - UNC Project, Lilongwe

REFERENCES:
- [Derived] Chen JS, Pettifor AE, Nelson JAE, Phiri S, Pasquale DK, Kumwenda W, Kamanga G, Cottrell ML, Sykes C, Kashuba ADM, Tegha G, Krysiak R, Thengolose I, Cohen MS, Hoffman IF, Miller WC, Rutstein SE. Brief Report: Blood and Genital Fluid Viral Load Trajectories Among Treated and Untreated Persons With Acute HIV Infection in Malawi. J Acquir Immune Defic Syndr. 2022 May 1;90(1):56-61. doi: 10.1097/QAI.0000000000002917. PMID 35044991
- [Derived] Dennis AM, Cohen MS, Rucinski KB, Rutstein SE, Powers KA, Pasquale DK, Phiri S, Hosseinipour MC, Kamanga G, Nsona D, Massa C, Hoffman IF, Pettifor AE, Miller WC. Human Immunodeficiency Virus (HIV)-1 Transmission Among Persons With Acute HIV-1 Infection in Malawi: Demographic, Behavioral, and Phylogenetic Relationships. Clin Infect Dis. 2019 Aug 16;69(5):853-860. doi: 10.1093/cid/ciy1006. PMID 30476007
- [Derived] Hino S, Grodensky C, Rutstein SE, Golin C, Smith MK, Christmas L, Miller W, Phiri S, Massa C, Kamanga G, Pettifor A. HIV status disclosure during acute HIV infection in Malawi. PLoS One. 2018 Jul 26;13(7):e0201265. doi: 10.1371/journal.pone.0201265. eCollection 2018. PMID 30048496

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through screening in two sexually transmitted disease clinics and two HIV testing sites in Lilongwe, Malawi.
Pre-assignment Details: Participants were evaluated in two stages: screening for acute HIV infection (AHI) and enrollment of persons with AHI for follow-up. As this is a pilot study, some outcomes refer to screening only. The original protocol called for 115 persons with AHI; only 46 persons were enrolled as the study period ended and funding expired.
Groups:
- Standard Counseling Arm: The SC arm consists of a single session of standard HIV prevention messages during HIV post-test counseling. The counseling will be comparable to that given to persons with established HIV infection with supplemental information regarding the acute stage of their infection.
  Standard HIV prevention messages: The standard counseling (SC) arm consists of a single session of standard HIV prevention messages during HIV post-test counseling. The counseling will be comparable to that given to persons with established HIV infection with supplemental information regarding the acute stage of their infection.
- Behavioral Intervention Arm: The BI arm consists of five counselor-delivered sessions based on the Information-Motivation-Behavioral Skills (IMB) Model. The sessions are designed to provide participants with the information, motivation, and skills needed to abstain or practice protected sex during the brief acute HIV period, as well as plan for long-term behavioral risk reduction.
  5 counselor-delivered sessions: The behavioral intervention (BI) arm consists of five counselor-delivered sessions based on the Information-Motivation-Behavioral Skills (IMB) Model. The sessions are designed to provide participants with the information, motivation, and skills needed to abstain or practice protected sex during the brief acute HIV period, as well as plan for long-term behavioral risk reduction.
- Behavioral Intervention Plus Antiretrovirals (BIA): The BIA arm consists of the same behavioral intervention plus antiretroviral drugs (ARVs) with raltegravir (400 mg twice daily) and fixed dose combination (FDC) emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) (200/300 mg daily) orally for 12 weeks.
  ARVs with raltegravir and emtricitabine/tenofovir disoproxil fumarate: The behavioral intervention and antiretroviral (BIA) arm consists of the same behavioral intervention plus antiretroviral drugs (ARV) with raltegravir (400mg twice daily) and fixed dose combination (FDC) emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) (200/300mg daily) orally for 12 weeks.
Period: Overall Study
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm | Behavioral Intervention Plus Antiretrovirals (BIA)
Started | 9 | 18 | 19
Completed | 9 | 18 | 19
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm | Behavioral Intervention Plus Antiretrovirals (BIA) | Total
Number analyzed (Participants) | 9 | 18 | 19 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (8.1) | 26.7 (5.1) | 27.1 (7.9) | 27.7 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 7 | 18
  Male | 5 | 11 | 12 | 28
Region of Enrollment [Number; unit: participants]
  Malawi | 9 | 18 | 19 | 46

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Persons Agreeing to be Screened for Acute HIV Infection Among Those Offered Screening
Time Frame: 1 year
Population: All persons screened
Measure: Number (95% Confidence Interval); unit: proportion of participants screened
Groups:
- Overall: All arms combined
Arm/Group | Overall
Number analyzed (Participants) | 14755
proportion of participants screened | 0.622 [0.614 to 0.630]

2. Primary Outcome: Prevalence of AHI Among Persons Screened
Description: Prevalence of AHI among all persons screened. This measure is among all persons screened, prior to randomization.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Overall
Number analyzed (Participants) | 9171
proportion of participants | 0.0073 [0.0057 to 0.0093]

3. Primary Outcome: Proportion of Persons With AHI Successfully Recruited Into the Study
Description: This outcome reflects the ability to recruit persons with AHI into a study. The outcome is based on the population prior to randomization.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: Proportion of persons with AHI recruited
Arm/Group | Overall
Number analyzed (Participants) | 67
Proportion of persons with AHI recruited | 0.69 [0.56 to 0.79]

4. Primary Outcome: Proportion of Participants Completing Full Course of ARVs in Arm BIA
Description: Proportion of participants in the BIA arm receiving full course of ARVs. This outcome is calculated among the BIA arm only, as that
Time Frame: 1 year
Population: Number of persons in BIA arm eligible for study-provided ARVs
Measure: Number (95% Confidence Interval); unit: proportion of BIA participants
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm | Behavioral Intervention Plus Antiretrovirals (BIA)
Number analyzed (Participants) | 0 | 0 | 12
proportion of BIA participants |  |  | 0.917 [0.615 to 0.998]

5. Primary Outcome: Proportion of Participants in Arm BI and BIA (Combined) Who Complete the 4 Behavioral Sessions Within 3 Weeks of Enrollment.
Description: In this pilot study, we addressed our ability to complete the behavioral intervention quickly. As two arms received the behavioral intervention, this outcome is combined across those two arms.
Time Frame: 1 year
Population: All persons in the two behavioral intervention arms
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Combined Behavioral Intervention Arms: Both the behavioral intervention and behavioral intervention plus antiretroviral arms are combined in this outcome
Arm/Group | Combined Behavioral Intervention Arms
Number analyzed (Participants) | 37
proportion of participants | 0.216 [0.098 to 0.382]

6. Primary Outcome: Proportion of Persons Completing All Scheduled Visits in Each Study Arm
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm | Behavioral Intervention Plus Antiretrovirals (BIA)
Number analyzed (Participants) | 9 | 18 | 19
Proportion of participants | 0.44 [0.14 to 0.79] | 0.44 [0.22 to 0.69] | 0.37 [0.16 to 0.62]

7. Primary Outcome: Number of Adverse Events
Description: Mean number of adverse events per group
Time Frame: one year
Measure: Mean (95% Confidence Interval); unit: number of events
Groups:
- Behavioral Intervention Plus ARV: The BIA arm:.
  Standard HIV prevention messages: A single session of standard HIV prevention messages during HIV post-test counseling with supplemental information regarding the acute stage of their infection.
  BI: Information-Motivation-Behavioral Skills Model: The behavioral intervention consists of five counselor-delivered sessions based on the Information-Motivation-Behavioral Skills (IMB) Model. The sessions are designed to provide participants with the information, motivation, and skills needed to abstain or practice protected sex during the brief acute HIV period, as well as plan for long-term behavioral risk reduction.
  Raltegravir: raltegravir (400 mg) administered orally twice daily for 12 weeks
  emtricitabine/tenofovir disoproxil fumarate: emtricitabine/tenofovir (200/300 mg daily) in a fixed dose combination administered orally for 12 weeks
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 9 | 18 | 19
number of events | 0.78 [0.31 to 1.6] | 1.3 [0.81 to 1.9] | 1.3 [0.85 to 1.9]

8. Secondary Outcome: Unprotected Sex Acts in Previous One Week - 12 Weeks
Description: The mean number of unprotected sex acts in previous one week, assessed at 12 weeks
Time Frame: 12 weeks
Population: Number includes enrolled persons who completed the ACASI interview within the window for this visit
Measure: Mean (95% Confidence Interval); unit: unprotected sex acts/week
Groups:
- Behavioral Intervention Plus ARV: The BIA arm:
  Standard HIV prevention messages: A single session of standard HIV prevention messages during HIV post-test counseling with supplemental information regarding the acute stage of their infection.
  BI: Information-Motivation-Behavioral Skills Model: The behavioral intervention consists of five counselor-delivered sessions based on the Information-Motivation-Behavioral Skills (IMB) Model. The sessions are designed to provide participants with the information, motivation, and skills needed to abstain or practice protected sex during the brief acute HIV period, as well as plan for long-term behavioral risk reduction.
  Raltegravir: raltegravir (400 mg) administered orally twice daily for 12 weeks
  emtricitabine/tenofovir disoproxil fumarate: emtricitabine/tenofovir (200/300 mg daily) in a fixed dose combination administered orally for 12 weeks
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 6 | 16 | 15
unprotected sex acts/week | 0 [0 to 0.6] | 0.5 [0.2 to 1.0] | 1.2 [0.7 to 1.9]

9. Secondary Outcome: Unprotected Sex Acts in Previous One Week - 26 Weeks
Description: The mean number of unprotected sex acts in previous one week, assessed at 26 weeks
Time Frame: 26 weeks
Population: Number includes enrolled persons who completed the ACASI interview within the window for this visit
Measure: Mean (95% Confidence Interval); unit: unprotected sex acts/week
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 8 | 14 | 15
unprotected sex acts/week | 0.25 [0.03 to 0.9] | 0.1 [0.02 to 0.5] | 0.5 [0.2 to 1.0]

10. Secondary Outcome: Unprotected Sex Acts in Previous One Week - 52 Weeks
Description: The mean number of unprotected sex acts in previous one week, assessed at 52 weeks
Time Frame: 52 weeks
Population: Number includes enrolled persons who completed the ACASI interview within the window for this visit
Measure: Mean (95% Confidence Interval); unit: unprotected sex acts/week
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 6 | 10 | 13
unprotected sex acts/week | 0.8 [0.3 to 1.9] | 0.2 [0.02 to 0.7] | 0 [0 to 0.3]

11. Secondary Outcome: Unprotected Sex Acts in Previous One Month - 12 Weeks
Description: The mean number of unprotected sex acts in previous one month, assessed at 12 weeks
Time Frame: 12 weeks
Population: Number includes enrolled persons who completed the ACASI interview within the window for this visit
Measure: Mean (95% Confidence Interval); unit: unprotected sex acts/month
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 6 | 16 | 15
unprotected sex acts/month | 0 [0 to 0.6] | 0.8 [0.4 to 1.4] | 0 [0 to 0.3]

12. Secondary Outcome: Unprotected Sex Acts in Previous One Month - 26 Weeks
Description: The mean number of unprotected sex acts in previous one month, assessed at 26 weeks
Time Frame: 26 weeks
Population: Number includes enrolled persons who completed the ACASI interview within the window for this visit
Measure: Mean (95% Confidence Interval); unit: unprotected sex acts/month
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 8 | 14 | 15
unprotected sex acts/month | 0.25 [0.03 to 0.9] | 0.2 [0.04 to 0.6] | 0.4 [0.1 to 0.9]

13. Secondary Outcome: Unprotected Sex Acts in Previous One Month - 52 Weeks
Description: The mean number of unprotected sex acts in previous one month, assessed at 52 weeks
Time Frame: 52 weeks
Population: Number includes enrolled persons who completed the ACASI interview within the window for this visit
Measure: Mean (95% Confidence Interval); unit: unprotected sex acts/month
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 6 | 10 | 13
unprotected sex acts/month | 0.8 [0.3 to 1.9] | 0.5 [0.2 to 1.2] | 0 [0 to 0.3]

14. Secondary Outcome: Cumulative Incidence of Gonorrhea, Chlamydial Infection and Trichomoniasis (Composite)
Description: Cumulative incidence, definied as at least one incident infection with either gonorrhea, chlamydia or trichomoniasis
Time Frame: 26 weeks
Population: Number includes all persons with gonorrhea, chlamydia, and trichomoniasis results who had not withdrawn from the study by the first scheduled STI tests
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 7 | 15 | 17
proportion of participants | 0.14 [0.004 to 0.58] | 0.33 [0.12 to 0.62] | 0.12 [0.015 to 0.36]

15. Secondary Outcome: Cumulative Incidence of Gonorrhea, Chlamydial Infection and Trichomoniasis (Composite)
Description: At least one incident infection with either gonorrhea, chlamydia or trichomoniasis
Time Frame: 52 weeks
Population: Number includes all persons with gonorrhea, chlamydia, and trichomoniasis results and who had at least one visit after Week 26
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 7 | 12 | 13
proportion of participants | 0.14 [0.004 to 0.58] | 0.42 [0.15 to 0.72] | 0.15 [0.019 to 0.45]

16. Secondary Outcome: Cumulative Incidence Herpes Simplex Virus Type 2
Description: cumulative incidence of herpes simplex virus type 2, assessed at 26 weeks. Persons with baseline positivity were excluded.
Time Frame: 26 weeks
Population: Number includes all persons who were confirmed HSV-2 negative at baseline and who had an informative test on or before Week 26
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 2 | 4 | 4
Proportion of participants | 0.5 [0.01 to 1] | 0.5 [0.07 to 0.9] | 0.25 [0.006 to 0.8]

17. Secondary Outcome: Cumulative Incidence Herpes Simplex Virus Type 2
Description: cumulative incidence of herpes simplex virus type 2, assessed at 52 weeks. Persons with baseline positivity were excluded.
Time Frame: 52 weeks
Population: Number includes all persons who were confirmed HSV-2 negative at baseline and who had an informative test on or before Week 52
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 2 | 3 | 3
Proportion of participants | 0.5 [0.01 to 1] | 1.0 [0.3 to 1.0] | 0.3 [0.008 to 0.9]

18. Secondary Outcome: Number of Partners Reporting for HIV Testing
Description: Number of partners per index reporting for HIV testing at any time during follow-up
Time Frame: 52 weeks
Measure: Mean (95% Confidence Interval); unit: partners per index participant
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 9 | 18 | 19
partners per index participant | 0.4 [0.1 to 1.1] | 0.4 [0.2 to 0.9] | 0.4 [0.1 to 0.8]

19. Secondary Outcome: Proportion of Partners Reporting for HIV Testing
Description: Proportion of sexual partners reporting for HIV testing among all sexual partners named by the index participants
Time Frame: 52 weeks
Population: The number of sexual partners named by the index participants is the denominator. For example, the 9 index participants in the standard arm named 35 partners. 4 partners presented, giving a proportion of 0.1 (4/35)
Measure: Number (95% Confidence Interval); unit: proportion of sex partners
Units Other Than Participants: sexual partners
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 9 | 18 | 19
Number analyzed (sexual partners) | 35 | 78 | 47
proportion of sex partners | 0.1 [0.03 to 0.3] | 0.1 [0.04 to 0.2] | 0.1 [0.01 to 0.3]

20. Secondary Outcome: Suppression of HIV RNA to <1000c/ml at 12 Weeks
Description: Proportion of persons in each arm with viral load <1000copies/ml at 12 weeks
Time Frame: 12 weeks
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 9 | 18 | 19
Proportion of participants | 0.5 [0.16 to 0.84] | 0.25 [0.07 to 0.52] | 0.72 [0.47 to 0.90]

21. Secondary Outcome: Time to HIV RNA Suppression <1000 c/ml
Description: median time to viral load suppression (<1000 c/ml)
Time Frame: From date of randomization until viral load suppression, up to 52 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 9 | 18 | 19
weeks | 39 [26 to 52] | 26 [26 to 39] | 16 [14 to 19]

22. Secondary Outcome: Blood HIV RNA Concentration at Week 12
Time Frame: 12 weeks
Population: Number includes enrolled persons who had an HIV RNA (blood) specimen available the window for this visit.
Measure: Median (Full Range); unit: copies/ml
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 6 | 16 | 15
copies/ml | 19411 [0 to 351974] | 22734 [20 to 741360] | 20 [0 to 2313294]

23. Secondary Outcome: Blood HIV RNA Concentration at Week 26
Time Frame: 26 weeks
Population: Number includes enrolled persons who had an HIV RNA (blood) specimen available the window for this visit.
Measure: Median (Full Range); unit: copies/ml
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 8 | 14 | 15
copies/ml | 8661 [0 to 208087] | 58504 [20 to 438579] | 6788 [0 to 196903]

24. Secondary Outcome: Blood HIV RNA Concentration at Week 52
Time Frame: 52 weeks
Population: Number includes enrolled persons who had an HIV RNA (blood) specimen available the window for this visit.
Measure: Median (Full Range); unit: copies/ml
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 6 | 10 | 11
copies/ml | 3248.5 [0 to 35668] | 6467.5 [0 to 432656] | 10876 [0 to 101615]

25. Secondary Outcome: Genital HIV RNA Concentration - Week 12, Women
Description: median HIV RNA concentration in cervical lavage fluid
Time Frame: 12 weeks
Population: Number includes enrolled women who had a genital HIV RNA sample obtained during the window for this visit.
Measure: Median (Full Range); unit: copies/ml
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 2 | 5 | 4
copies/ml | 82.5 [0 to 165] | 0 [0 to 6501] | 38.5 [0 to 90]

26. Secondary Outcome: Genital HIV RNA Concentration - Week 26, Women
Description: median HIV RNA concentration in cervical lavage fluid
Time Frame: 26 weeks
Population: Number includes enrolled women who had a genital HIV RNA sample obtained during the window for this visit.
Measure: Median (Full Range); unit: copies/ml
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 4 | 4 | 3
copies/ml | 11.5 [0 to 564] | 0 [0 to 92] | 164 [0 to 2500]

27. Secondary Outcome: Genital HIV RNA Concentration - Week 52, Women
Description: median HIV RNA concentration in cervical lavage fluid
Time Frame: 52 weeks
Population: Number includes enrolled women who had a genital HIV RNA sample obtained during the window for this visit.
Measure: Median (Full Range); unit: copies/ml
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 3 | 2 | 2
copies/ml | 0 [0 to 124] | 219 [0 to 438] | 2111 [350 to 3872]

28. Secondary Outcome: Genital HIV RNA Concentration - Week 12, Men
Description: median HIV RNA concentration as measured in semen
Time Frame: 12 weeks
Population: Number includes enrolled men who had a genital HIV RNA sample obtained during the window for this visit.
Measure: Median (Full Range); unit: copies/ml
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 2 | 5 | 7
copies/ml | 25364 [1636 to 49092] | 446 [0 to 23798] | 0 [0 to 782]

29. Secondary Outcome: Genital HIV RNA Concentration - Week 26, Men
Description: median HIV RNA concentration as measured in semen
Time Frame: 26 weeks
Population: Number includes enrolled men who had a genital HIV RNA sample obtained during the window for this visit.
Measure: Median (Full Range); unit: copies/ml
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 2 | 3 | 4
copies/ml | 9456 [788 to 18124] | 292 [0 to 2024] | 0 [0 to 0]

30. Secondary Outcome: Genital HIV RNA Concentration - Week 52, Men
Description: median HIV RNA concentration as measured in semen
Time Frame: 52 weeks
Population: Number includes enrolled men who had a genital HIV RNA sample obtained during the window for this visit.
Measure: Median (Full Range); unit: copies/ml
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm Only | Behavioral Intervention Plus ARV
Number analyzed (Participants) | 1 | 2 | 5
copies/ml | 13088 [13088 to 13088] | 66 [0 to 132] | 0 [0 to 826]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Standard Counseling Arm | Behavioral Intervention Arm | Behavioral Intervention Plus Antiretrovirals (BIA)
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 4/9 | 11/18 | 13/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Counseling Arm (N=9) | Behavioral Intervention Arm (N=18) | Behavioral Intervention Plus Antiretrovirals (BIA) (N=19)
genital discharge/sores (Reproductive system and breast disorders) | 0 (0) | 3 (4) | 4 (4)
fever/chills (General disorders) | 2 (2) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0
Numbness (feet) (Nervous system disorders) | 0 | 0 | 1 (2)
finger nail changes (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0
headache (General disorders) | 0 | 2 (2) | 1 (1)
nausea/vomiting/diarrhea/abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (5) | 6 (10)
Skin rash/skin sores/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (7) | 3 (3)
toothache (Gastrointestinal disorders) | 0 | 0 | 1 (1)
weakness (General disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Please note that this trial was a pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No